CLINICAL TRIAL: NCT01716013
Title: A Multi-Center, Prospective, Open-label, Randomized Study of the Safety and Efficacy of BondEase™ Topical Skin Adhesive for the Closure of Traumatic Lacerations and Surgical Incisions
Brief Title: Safety and Efficacy Study of BondEase to Treat Traumatic Lacerations and Surgical Incisions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: OptMed, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PD-100-002
Record Dates: First submitted 2012-10-21; First posted 2012-10-29 (Estimated); Results first posted 2016-11-18 (Estimated); Last update posted 2017-01-09 (Estimated); Status verified 2016-11

CONDITIONS: Traumatic Lacerations or Surgical Incisions
MeSH Terms: conditions — Surgical Wound

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- BondEase (Experimental): Topical Skin Adhesive
  Interventions: Device: BondEase
- CWCD (Active Comparator): Conventional Wound Closure Devices (CWCD) including: sutures, staples, or adhesive strips
  Interventions: Procedure: CWCD

INTERVENTIONS:
Device: BondEase — topical skin adhesive
  Arms: BondEase
Procedure: CWCD — traditional closure methods of sutures, staples or adhesive strips
  Arms: CWCD

SUMMARY:
To demonstrate that BondEase™ and conventional wound closure devices (CWCD) are the same in terms of cosmesis (appearance) of the repaired wound when these devices are used for closure of surgical and traumatic wounds .

To demonstrate safety of BondEase™.

DETAILED DESCRIPTION:
This is a two-phase, multi-center, prospective, randomized, parallel-group study, in which a total of 153 subjects (102 in the BondEase™ group and 51 in the CWCD group) with traumatic lacerations and incisions will be enrolled. Overall, eligible subjects will be randomized in a pre-defined 2:1 ratio to BondEase™ skin adhesive or CWCD.

In Part 1 of the study 30 subjects will be randomized in a 2:1 ratio (BondEase™ : CWCD). This part of the study is designed to assess the feasibility and validate use of the device. Pediatric subjects younger than age 18 will not be included in this part of the trial. The results from these 30 subjects will be compiled and submitted to FDA for review and approval prior to proceeding with Part 2. Part 2 of the study will only be initiated after FDA indicates it is acceptable to begin. In Part 2 of the study a total of 123 subjects will be randomized, of which 82 subjects will be randomized to the BondEase™ group and 41 subjects to the CWCD group. This will result in 102 subjects in the BondEase™ group and 51 subjects in the CWCD group across the both parts of the trial.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects at least 1 year of age (for Part 2 only) or at least 18 years of age (for both Part 1 and Part 2).
2. Has a wound requiring surgical repair, where the use of a tissue adhesive is appropriate
3. Is in good general health
4. Subject or the guardian understands and is willing to sign informed consent prior to study entry and agrees to be available for the Day 10, Day 28, and Day 90 (Part 1/pilot phase only) follow-up visits

Exclusion Criteria:

1. Significant or multiple traumas
2. Known peripheral vascular disease
3. Known diabetes mellitus type 1 or type 2
4. Known blood clotting disorder
5. Patient or family history of keloid formation or hypertrophy
6. Known HIV seropositivity or is immunocompromised
7. Been treated with an investigational drug or medical device in the past 30 days
8. A hypersensitivity or contraindication to any of the components of BondEase™
9. Known pre-operative systemic or local infection
10. Any other diseases or conditions which might interfere with the wound healing process
11. The wound to be treated with the test device may not have any of the following characteristics:

    * A "burst" or stellate laceration
    * Heavily contaminated (Contaminated Wound: wounds that are grossly contaminated with foreign material requiring extensive cleansing.
    * Human or animal bite
    * Decubitus etiology
    * Evidence of active infection or gangrene
    * On mucosal surfaces or across mucocutaneous junctions (e.g., oral cavity, lips)
    * On an area which may be regularly exposed to body fluids or with dense natural hair, (e.g., scalp)
    * Under tension or over a joint

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Actual)
Dates: Start 2012-09; Primary Completion 2014-01 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Orlando Regional Medical Center, Orlando, Florida
  - Northwestern University, Chicago, Illinois
  - DC Cosmetics, Chevy Chase, Maryland
  - Albany Medical Center, Albany, New York
  - Sadick Research Group, New York, New York
  - Wake Forest Baptist Health, Wake Forest, North Carolina

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | BondEase | CWCD
Started | 108 | 54
Completed | 105 | 54
Not Completed | 3 | 0

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population
Groups:
- Total: Total of all reporting groups
Arm/Group | BondEase | CWCD | Total
Number analyzed (Participants) | 105 | 54 | 159
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.4 (23.1) | 47.7 (22.3) | 45.5 (22.8)
Gender [Count of Participants; unit: Participants]
  Female | 49 | 24 | 73
  Male | 56 | 30 | 86
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 21 | 5 | 26
  Not Hispanic or Latino | 84 | 49 | 133
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 16 | 7 | 23
  White | 83 | 46 | 129
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 4 | 0 | 4
Wound type [Number; unit: participants]
  Injury (Laceration) | 27 | 13 | 40
  Surgical incision | 78 | 41 | 119

OUTCOME MEASURES:

1. Primary Outcome: 100% Wound Apposition at 10 Days
Description: Percentage of subjects in whom 100% wound edge apposition is achieved at 10 days (±3 days) post-procedure.
Time Frame: 10 days
Population: Per protocol population (primary analysis dataset)
Measure: Number; unit: percentage of participants
Arm/Group | BondEase | CWCD
Number analyzed (Participants) | 96 | 51
percentage of participants | 77.1 | 80.4

2. Secondary Outcome: Optimal Cosmetic Outcome at 28 Days (Score of 6)
Description: Incidence of wounds with an optimal cosmetic outcome (score of 6) at 28 days.
  One point was scored for the absence of, and no point was scored for the presence of, any of the following six items:
  * Stepoff of borders (edges not on the same plane)
  * Contour irregularities (wrinkled skin near wound)
  * Margin separation (gap between sides)
  * Edge inversion (wound not properly everted)
  * Excessive distortion (swelling or edema or infection)
  * Poor overall appearance.
  The overall cosmesis score was determined by adding the scores of each individual item. An overall score of six was considered an optimal score outcome. Any score below six was considered suboptimal.
Time Frame: 28 days
Population: Intent-to-treat (ITT) population
Measure: Number; unit: percentage of participants
Arm/Group | BondEase | CWCD
Number analyzed (Participants) | 105 | 54
percentage of participants | 70.5 | 64.8

3. Secondary Outcome: ≥ 50% Wound Apposition at 10 Days
Description: Incidence of wounds ≥50% apposed (10 ± 3 days)
Time Frame: 10 days
Population: Intent-to-treat (ITT) population
Measure: Number; unit: percentage of participants
Arm/Group | BondEase | CWCD
Number analyzed (Participants) | 105 | 54
percentage of participants | 93.3 | 96.3

4. Other Pre Specified Outcome: Wound Dehiscence Requiring Treatment
Description: Wound dehiscence requiring treatment; i.e., need for supplemental closure due to dehiscence at any time, from closure through follow-up
Time Frame: 28 Days and 90 days
Population: Intent-to-Treat (ITT) population
Measure: Number; unit: percentage of participants
Arm/Group | BondEase | CWCD
Number analyzed (Participants) | 105 | 54
percentage of participants | 0 | 0

ADVERSE EVENTS:
Arm/Group | BondEase | CWCD
Serious Adverse Events (participants affected / at risk) | 0/105 | 0/54
Other Adverse Events (participants affected / at risk) | 14/105 | 6/54
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BondEase (N=105) | CWCD (N=54)
Dehiscence with No Need for Retreatment (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Mild Scar (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 7 (7) | 4 (4) — Acute Inflammation at 10 days
Edema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Acute Inflammation at 10 days
Pain (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2) — Acute Inflammation at 10 days

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor shall have been furnished copies of any proposed publication or presentation at least thirty (30) days in advance of the submission of such proposed publication or presentation to a journal, editor, or other third party. Sponsor reserves the right to object to the proposed presentation or publication.